CLINICAL TRIAL: NCT05631470
Title: Diagnostic Accuracy for Hemodynamical Intracranial Atherosclerotic Diseases (ICAS) of Magnetic-Resonance-based Fractional Flow Reserve (MR-FFR) Comparing With Pressure-wire-based FFR.
Brief Title: Diagnostic Accuracy for Hemodynamically ICAS of MR-FFR Comparing With Pressure-wire-based FFR.
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: National Key Research and Development Project, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: XWFFR-2
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-01

CONDITIONS: Stroke, Ischemic; Intracranial Atherosclerosis
Keywords: Intracranial atherosclerotic diseases; Fractional Flow Reserve
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled: Participants with ICAS will be scheduled for both MR screening and pressure-wire-based FFR measurement.
  Interventions: Diagnostic Test: MR screening

INTERVENTIONS:
Diagnostic Test: MR screening — This study is to compare the results of MR-FFR with pressure-wired-based FFR measurement.
  Other Names: Pressure-wire-based FFR

SUMMARY:
The aim of this study was to determine the diagnostic accuracy of MR-FFR to detect functionally significant ICAS comparing with pressure-wire-based FFR.

DETAILED DESCRIPTION:
This study will perform a head-to-head comparison between MR-FFR and pressure-wire-based FFR in patients with ICAS. Pressure-wire-based FFR will be used as the gold standard for intravascular pressure gradient measurement. The efficacy and safety of non-invasive FFR will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older.
2. Patients with transient ischemic attack (TIA) or nondisabling ischemic stroke caused by a focal ICAS lesion located in intracranial anterior circulation (intracranial internal carotid artery and their major branches).
3. 50% to 99% stenosis (calculated by modified WASID method) of responsible arterial occlusion, confirmed by digital subtraction angiography (DSA).
4. Informed of the study protocol and objectives.

Exclusion Criteria:

1. Non-atherosclerotic MCA stenosis
2. Combined with moderate or severe stenosis of other extracranial and intracranial arteries
3. Previous endovascular treatment or surgery for cerebrovascular diseases
4. Large cerebral infarction (more than 1/2 MCA perfusion area)
5. Combined with other neurological diseases, such as aneurysm, arteriovenous malformation, tumor, hydrocephalus, cerebral trauma, cerebral hemorrhage, multiple sclerosis, epilepsy and intracranial infection.
6. Vascular abnormality or stunting, resulting in the impossibility of endovascular intervention
7. Liver and kidney dysfunction, or severe allergy to the contrast agent
8. Severe coagulation dysfunction
9. Pregnancy or in the preparation for pregnancy
10. Patients who cannot tolerate or do not allow MR screening, including metal implanting and claustrophobia
11. Patients with severe dementia or mental disorders, who cannot cooperate with examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic ICAS resorting to endovascular therapy in our center were recruited consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of MR-FFR measurement. | 3 days
  The consistency of the two groups in the interpretation of hemodynamic conditions across the ICAS lesion.

SECONDARY OUTCOMES:
The rate of all-cause stroke and mortality. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China